CLINICAL TRIAL: NCT06086652
Title: Role of Positron Emission Tomography in Detecting Primary Tumor in Cases of Metastases of Unknown Origin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doaa Ibrahim Mohamed, lecturer of nuclear medicine, faculty of medicine, Sohag university, Sohag University
Other Study IDs: Soh-Med-23-09-2PD
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Metastasis of Unknown Origin
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT — detection of possible primary tumor

SUMMARY:
In most cases of malignancies, the site of origin of the cancer is clear at presentation or identified soon after. However, Metastatic cancer of unknown primary site (MUO) accounts for 3-5% of all malignant neoplasms, and it is defined as metastatic cancer from an unknown primary site, for which no original site can be detected even after performing all possible tests. Most common metastatic sites include the liver, lymph nodes, lungs, and bones.

18F-fluoro-2-deoxyglucose positron emission tomography (FDG-PET) allows whole-body tumor detection and has proven to be useful in patients with metastasis of unknown primary tumor.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years Patients with metastatic tumor. Primary site was not detected with other radiological examinations Both male and female.

Exclusion Criteria:

Patients with known primary tumor Pregnancy. Age < 18 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Age > 18 years Patients with metastatic tumor. Primary site was not detected with other radiological examinations Both male and female.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
primary tumor for metastasis of unknown origin | one month
  primary tumor for metastasis of unknown origin

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Strate I, Kazemzadeh F, Nagtegaal ID, Robbrecht D, van de Wouw A, Padilla CS, Duijts S, Esteller M, Greco FA, Pavlidis N, Qaseem A, Snaebjornsson P, van Zanten SV, Loef C. International consensus on the initial diagnostic workup of cancer of unknown primary. Crit Rev Oncol Hematol. 2023 Jan;181:103868. doi: 10.1016/j.critrevonc.2022.103868. Epub 2022 Nov 23. PMID 36435296
- [Background] Kwee TC, Kwee RM. Combined FDG-PET/CT for the detection of unknown primary tumors: systematic review and meta-analysis. Eur Radiol. 2009 Mar;19(3):731-44. doi: 10.1007/s00330-008-1194-4. Epub 2008 Oct 17. PMID 18925401